CLINICAL TRIAL: NCT06226935
Title: Comparative Analysis of Glaucoma Screening Uptake Among First-Degree Relatives in Community-Based and Hospital-Based Approaches
Status: Completed | Type: Observational
Sponsor: Phrapokklao Hospital,Thailand (Other)
Responsible Party: Principal Investigator, Porntip Nitikarun, ophthalmology department, Phrapokklao Hospital,Thailand
Other Study IDs: Phrapokklao Hospital
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Evaluate the Differences in Glaucoma Screening Uptake Among FDRs in Community and Hospital-based
Keywords: Glaucoma Screening; First-Degree Relatives; Community-Based Approach; Hospital-Based Approach; Familial Risk Factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In conclusion, the study shows that the hospital-based group had a significantly higher screening uptake than the community-based group, reflecting that information from ophthalmologists and registered ophthalmic nurses is more effective and well-received than that from village health volunteers. The study suggests that increasing education and support for village health volunteers could enhance screening uptake. Factors influencing uptake include the age of FDRs, place of residence, education, presenting VA of probands, and treatment of probands. Utilizing this study's findings, spreading knowledge and training health officials at the district and sub-district levels could increase understanding of glaucoma and improve communication with the general public and at-risk groups, potentially increasing the response rate. Additionally, implementing a national free screening glaucoma program for at-risk populations, both in and outside hospitals, and organizing mobile screening units at the district level could be an effective prevention strategy against permanent vision loss from glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* All patients with POAG who had a treatment history in the ophthalmology outpatient department of Prapokklao Hospital, Chanthaburi Province, were identified from the Electronic Medical Record (EMR) database with the 10th revision of the International Statistical Classification of Diseases and Related Health Problems (ICD-10) " Primary open angle glaucoma H40.1" between 1 january 2022 to 31 october 2022. A total of 1304 patients were included in this study.

Exclusion Criteria:

* Excluding those with closed-angle glaucoma and secondary glaucoma due to other conditions such as accidents, post-surgical complications, uveitis, or congenital.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: These probands were then divided into two non-randomized groups: The first group, hospital-based, included all probands receiving treatment in the ophthalmology outpatient department from 1 dec 2022 to 28 feb 2023. These patients received information about glaucoma from ophthalmologists and registered ophthalmic nurses, along with a brochure.
  These patients were asked to invite FDRs-parents, siblings, and offspring aged 40 years and above - to participate screening.
  The second group, community-based, involved randomly selecting districts in Chanthaburi In this group, village health volunteers trained in glaucoma knowledge by ophthalmologists distributed brochures and educated patients and FDRs, similar to the hospital-based group. These FDRs were then invited to participate in the glaucoma screening program one month later, with ophthalmologists at health stations near homes in Muang district and Laem Sing Hospital between 1 mar 2023 to 31 may 2023.
Sampling Method: Non-Probability Sample
Enrollment: 1304 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
This study aimed to evaluate the differences in glaucoma screening uptake among FDRs in community and hospital-based settings | Jan 1,2022-May 31,2023
  All patients with POAG who had a treatment history in OPD of Prapokklao Hospital, Chanthaburi Province, were identified from EMR database with ICD-10 "H40.1". These probands were then divided into two non-randomized groups: The first group, hospital-based, these patients received information from ophthalmologists and registered ophthalmic nurses, along with a brochure .Subsequently, these patients were asked to invite their FDRs - aged 40 years and above - to participate in screening. The second group, community-based, involved randomly selecting districts in Chanthaburi Province for screening, including Muang and Laem Sing districts. After excluded the patients already participating in the hospital-based group from the EMR database, 682 probands remained in the second group. In this group, village health volunteers trained in glaucoma knowledge by ophthalmologists distributed brochures and educated patients and FDRs.

SECONDARY OUTCOMES:
This study investigated the determinants influencing participation in glaucoma screening programs and the prevalence of glaucoma in FDRs. | Jan 1,2022-May 31,2023
  All glaucoma patients and their FDRs underwent a detailed by history taking information such as age, underlying disease, address, time of diagnosis glaucoma, medical history treatment of glaucoma and relationship with the glaucoma patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Phrapokklao Hospital, Chanthaburi, Thailand